CLINICAL TRIAL: NCT03465033
Title: Early Physiotherapy, Mandibular Motion and Sensorial Recovery After Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Rafael Martínez-Conde Llamosas, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10_2017_194
Record Dates: First submitted 2018-02-11; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Mandibular Range of Motion; Pain; Sensorial Disturbance
Keywords: Orthognathic surgery; Jaw rehabilitation; Jaw Physiotherapy; Pain; Mandibular range of motion; Sensorial disturbance
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Patients undergoing OS will be studied. All patients will be told that two interventions are compared but they will not know which one is the usual care or the early physiotherapy. All of them will receive instructions of basic care after surgery: use of intermaxillary elastics, soft diet during the first month and semi-soft during the second month. Patients will be asked to remove the intermaxillary elastics 30min before the measurements.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All patients will be told that two interventions are compared but they will not know which one is the usual care or the early physiotherapy. Professionals that will evaluate the measurements and the investigators that will make the statistical analysis, all will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients will receive basic indications of rehabilitation consisting of daily mobilization of the jaw (perform several movements a day opening movements, laterotrusion and mouth protrusion).
- Early Physiotherapy (Experimental)
  Interventions: Other: Early Physiotherapy

INTERVENTIONS:
Other: Early Physiotherapy — From T1 to T2 patients will perform 3 daily repetitions of active exercises:1 5 repetitions of oral opening exercises and bilateral manual progressive stretching, protrusion and maximum lateralization of the jaw on both sides, holding each movement for 5s and a session of cryotherapy applied to the masseter, temporal and suprahyoid muscles for 120s in two 60s sessions. They will also perform 30 repetitions of exercises aimed at improving the labial seal (inflate cheeks) and the symmetry of the upper lip (broad smile). From T2 to T3 30 repetitions of the same exercises will be performed and passive progressive opening will be implemented by "clamping" Patients will also perform isometric contraction exercises in opening, closing, laterotrusion, protrusion and retrusion. Each movement will be repeated 5 times and it will remain for 5s.
  Arms: Early Physiotherapy

SUMMARY:
Several studies describe that the maximum mandibular opening decreases 60% -70% immediately after orthognathic surgery (OS) and other variables, including laterotrusion, movement speed and facial mimic also decrease drastically. In addition, patients frequently experience temporary or permanent sensory orofacial disturbances ranging from 9% to 76% of cases.

It has been described that scheduled early physiotherapy reduces these complications.

DETAILED DESCRIPTION:
Before the surgical intervention (T0) the maximum interincisal oral opening measurement, laterotrusion and maximum protrusion will be recorded by digital caliber. The overbite and the overjet, length of upper lip and lower facial third will be measured. The symmetry of the upper lip in a forced smile will be determined. The measurements made at T0 will be repeated at T1 (2 weeks after surgery), T2 (5 weeks after surgery), T3 (9 weeks after surgery), T4 (12 weeks after surgery), T5 (24 weeks after surgery) and T6 (after orthodontic removal).The level of pain during the measurements of the mandibular movements will be recorded in the Visual Analogue Scale, and the self-reported area of the orofacial sensory alterations by means of a diagram and the objective area by means of the sensory discrimination test of two points will be determined. In T4, the impact of the status of the function and oral structures on daily activities will be recorded through a self-pass questionnaire based on the Oral Index Daily Performance questionnaire (OIDP-sp). In the T6 the measurement of laterotrusion, protrusion and retrusion movements measured by Gysi Gothic arch will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Patients treated with orthodontics and OS for correction of dentofacial deformities.

Exclusion Criteria:

* Patients diagnosed with temporomandibular disorders
* Patients diagnosed with orofacial pain
* Patients diagnosed with orofacial sensory alterations
* Patients not treated with orthodontics
* Patients and who need to undergo OS interventions for the treatment of Sleep Apnea-Hypopnea Syndrome
* Patients that present cleft palate
* Patients that present cleft lip
* Patients diagnosed with syndromes that affect the orofacial structures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2020-03-09 (Estimated); Study Completion 2021-03-12 (Estimated)

PRIMARY OUTCOMES:
Pain during mandibular movements | week 12 (T4)
  The level of pain during the measurements of the mandibular movements will be registered using a Visual Analogue Scale, in which point 0 represents "no pain" and point 10 "maximum pain". Values under point 5 are considered to represent mild pain and values above point 5 severe pain
Maximum interincisor opening | week 12 (T4)
  The maximum interincisal oral opening measurement will be recorded by digital caliber

SECONDARY OUTCOMES:
Lip symmetry | Before OS (T0), week 2 after surgery (T1), week 5 (T2), week 9 (T3), week 12 (T4), week 24 (T5), and after orthodontic removal: up to one year after OS (T6)
  Lip symmetry will be recorded by facial photography of the patient in broad smile
Orofacial sensitivity | Week 2 after surgery (T1), week 5 (T2), week 9 (T3), week 12 (T4), week 24 (T5), and after orthodontic removal: up to one year after OS (T6)
  Self-reported area of orofacial sensory alterations will be measured by means of a diagram and the objective area by means of the sensory discrimination test of two points.
Laterotrusion | Before OS (T0), week 2 after surgery (T1), week 5 (T2), week 9 (T3), week 12 (T4), week 24 (T5), and after orthodontic removal: up to one year after OS (T6)
  The oral laterotrusion measurement will be recorded by digital caliber
Protrusion | Before OS (T0), week 2 after surgery (T1), week 5 (T2), week 9 (T3), week 12 (T4), week 24 (T5), and after orthodontic removal: up to one year after OS (T6)
  The oral protrusion measurement will be recorded by digital caliber
Impact of the status of the oral function and structures on daily activities | Week 12 (T4)
  The impact of the status of the oral function and structures on daily activities will be recorded through a self-pass questionnaire based on the Oral Index Daily Performance questionnaire (OIDP-sp)). In the OIDP index impacts are quantified by multiplying the frequency and severity scores to obtain the performance score for each of eight dimensions (eating, speaking, cleaning teeth, working, social relation, sleeping/relaxing, smiling and emotional status). The sum of these scores is considered the total impact score. This total score is divided by the maximum possible score and multiplied by 100 to give the percentage score. This scoring system yields an intuitive oral impact score.
Functional oral movements - Gysi Gothic arch | After orthodontic removal: up to one year after OS (T6)
  The measurement of laterotrusion, protrusion and retrusion movements measured by Gysi Gothic arch will be performed and the functional oral movements capacity will be measured bay the total of millimeters of all movements

CONTACTS AND LOCATIONS:
Locations (1):
- Department fo Stomatology II, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altmann EB. Myofunctional therapy and orthognathic surgery. Int J Orofacial Myology. 1987 Nov;13(3):2-12. No abstract available. PMID 3479402
- [Background] Bell WH, Gonyea W, Finn RA, Storum KA, Johnston C, Throckmorton GS. Muscular rehabilitation after orthognathic surgery. Oral Surg Oral Med Oral Pathol. 1983 Sep;56(3):229-35. doi: 10.1016/0030-4220(83)90001-4. PMID 6579456
- [Background] Bonine FL. Exercises to improve facial animation after orthognathic surgery. J Oral Maxillofac Surg. 1998 Feb;56(2):281. doi: 10.1016/s0278-2391(98)90898-9. No abstract available. PMID 9461161
- [Background] Dietrich EM, Griessinger N, Neukam FW, Schlittenbauer T. Consultation with a specialized pain clinic reduces pain after oral and maxillofacial surgery. J Craniomaxillofac Surg. 2017 Feb;45(2):281-289. doi: 10.1016/j.jcms.2016.12.009. Epub 2016 Dec 14. PMID 28057402
- [Background] Essick GK, Phillips C, Kim SH, Zuniga J. Sensory retraining following orthognathic surgery: effect on threshold measures of sensory function. J Oral Rehabil. 2009 Jun;36(6):415-26. doi: 10.1111/j.1365-2842.2009.01954.x. Epub 2009 Apr 28. PMID 19422435
- [Background] Gallerano G, Ruoppolo G, Silvestri A. Myofunctional and speech rehabilitation after orthodontic-surgical treatment of dento-maxillofacial dysgnathia. Prog Orthod. 2012 May;13(1):57-68. doi: 10.1016/j.pio.2011.08.002. Epub 2012 Jan 25. PMID 22583588
- [Background] Hong SO, Baek SH, Choi JY. Physical Therapy for Smile Improvement After Orthognathic Surgery. J Craniofac Surg. 2017 Mar;28(2):422-426. doi: 10.1097/SCS.0000000000003099. PMID 28114219
- [Background] Montero J, Bravo M, Albaladejo A. Validation of two complementary oral-health related quality of life indicators (OIDP and OSS 0-10 ) in two qualitatively distinct samples of the Spanish population. Health Qual Life Outcomes. 2008 Nov 18;6:101. doi: 10.1186/1477-7525-6-101. PMID 19019208
- [Background] Phillips C, Kim SH, Tucker M, Turvey TA. Sensory retraining: burden in daily life related to altered sensation after orthognathic surgery, a randomized clinical trial. Orthod Craniofac Res. 2010 Aug;13(3):169-78. doi: 10.1111/j.1601-6343.2010.01493.x. PMID 20618719
- [Background] Teng TT, Ko EW, Huang CS, Chen YR. The Effect of early physiotherapy on the recovery of mandibular function after orthognathic surgery for Class III correction: part I--jaw-motion analysis. J Craniomaxillofac Surg. 2015 Jan;43(1):131-7. doi: 10.1016/j.jcms.2014.10.025. Epub 2014 Nov 1. PMID 25439086